CLINICAL TRIAL: NCT07311109
Title: A Prospective, Single-center, Randomized Controlled Clinical Study Evaluating the Efficacy and Safety of Hyperbaric Oxygen Therapy as an Adjunctive Treatment for Chronic Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, Chief, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0202502
Record Dates: First submitted 2025-12-09; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-10

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: chronic heart failure; HBOT
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen therapy (Experimental): Participants in the control arm will receive guideline-directed medical therapy exclusively, founded on the "New Four Pillars" regimen (ARNI/ACEI/ARB + Beta-blocker + MRA + SGLT2 inhibitor) for chronic heart failure.
  The hyperbaric oxygen therapy protocol consists of 3 treatment courses, with each course comprising 10 sessions. There is a one-month interval between each course.
  The therapy is administered in a multi-place chamber at a pressure of 0.2 MPa (2 ATA). The treatment protocol per session is as follows: 20 minutes of compression, followed by two 30-minute periods of oxygen inhalation via mask, separated by a 10-minute air break, and finally 20 minutes of decompression. The total duration per session is 110 minutes.
  Sessions are conducted 5 times per week, making the total duration of each treatment course 14 days.
  Interventions: Other: hyperbaric oxygen therapy
- standard guideline-directed medical therapy for chronic heart failure (Sham Comparator): Participants in the control arm will receive guideline-directed medical therapy exclusively, founded on the "New Four Pillars" regimen (ARNI/ACEI/ARB + Beta-blocker + MRA + SGLT2 inhibitor) for chronic heart failure. Apart from the absence of hyperbaric oxygen therapy, all other management strategies are consistent with those in the experimental arm.
  Interventions: Other: hyperbaric oxygen therapy

INTERVENTIONS:
Other: hyperbaric oxygen therapy — The therapy is administered in a multi-place chamber at a pressure of 0.2 MPa (2 ATA). The treatment protocol per session is as follows: 20 minutes of compression, followed by two 30-minute periods of oxygen inhalation via mask, separated by a 10-minute air break, and finally 20 minutes of decompression. The total duration per session is 110 minutes.

SUMMARY:
This study aims to investigate whether adjunctive hyperbaric oxygen therapy, compared to guideline-directed medical therapy with the "New Four Pillars" (ARNI/ACEI/ARB + β-blocker + MRA + SGLT2 inhibitor) alone, improves cardiac function in patients with chronic heart failure, and to evaluate its efficacy and safety.

DETAILED DESCRIPTION:
1. Study Design This is a prospective, single-center, randomized controlled clinical trial designed to evaluate the efficacy and safety of hyperbaric oxygen therapy as an adjunctive treatment for chronic heart failure.
2. Randomization After confirming eligibility, participants will be randomized in a 1:1 ratio via a web-based randomization system into either the experimental group (hyperbaric oxygen therapy plus standard medication) or the control group (standard medication alone).
3. Treatment Protocol Patients diagnosed with chronic heart failure at the center, who meet the criteria and have no absolute contraindications for hyperbaric oxygen therapy, will be enrolled. Specifically, the study will enroll patients with Heart Failure with Reduced Ejection Fraction (HFrEF, EF ≤40%) as per the latest guidelines.

   Experimental Group: Participants will receive hyperbaric oxygen therapy in addition to stable, guideline-directed medical therapy based on the "New Four Pillars" (ARNI/ACEI/ARB + Beta-blocker + MRA + SGLT2 inhibitor).

   Control Group: Participants will receive only the standard guideline-directed medical therapy ("New Four Pillars" as above) for chronic heart failure. All other aspects of care are identical to the experimental group, except for the hyperbaric oxygen therapy.

   Given that chronic heart failure requires long-term management, the hyperbaric oxygen protocol is divided into three courses to consolidate and maintain efficacy, as well as to improve patients' oxygen reserve capacity and tolerance. Each course consists of 10 sessions, with a one-month interval between courses.

   The hyperbaric oxygen treatment will be administered in a multi-place chamber at a pressure of 0.2 MPa (2 ATA). The session protocol is as follows: 20 minutes of compression, followed by two 30-minute periods of oxygen inhalation via mask, separated by a 10-minute air break, and finally 20 minutes of decompression. The total duration per session is 110 minutes. Sessions are conducted 5 times per week, making the total duration of each treatment course 14 days.
4. Follow-up After randomization and initiation of treatment, clinical follow-up visits will be conducted to collect data. For the experimental group, follow-ups will occur one day after the completion of each hyperbaric oxygen course. All participants (both groups) will undergo additional follow-ups at 3 months, 6 months, and 12 months after the complete hyperbaric oxygen treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic Criteria

   Diagnosis of chronic heart failure according to the Chinese Guidelines for the Diagnosis and Management of Heart Failure (2024), and meeting the following conditions:

   1.1 Left Ventricular Ejection Fraction (LVEF) ≤ 40% (HFrEF group). 1.2 Presence of chronic HF symptoms (NYHA functional class II-IV) or objective evidence (e.g., elevated natriuretic peptides, structural cardiac abnormalities).

   1.3 Disease duration ≥ 3 months, with no adjustments to the foundational anti-heart failure regimen within the past month.
2. Age and Informed Consent 2.1 Aged 18 to 70 years (inclusive). 2.2 Understand the study purpose and provide signed informed consent.
3. Treatment Stability 3.1 Received guideline-recommended, standardized "New Four Pillars" anti-heart failure therapy (ARNI/ACEI/ARB + β-blocker + MRA + SGLT2 inhibitor) for at least 2 weeks prior to enrollment, with no changes in the past month.

3.2 No diuretic dose adjustments within the past 5 days and no clinical signs of fluid overload (e.g., weight gain of ≥ 2 kg/week, new-onset pulmonary edema).

-

Exclusion Criteria:

* Absolute Contraindications

  1. Untreated pneumothorax or pneumomediastinum.
  2. Claustrophobia, agitation or inability to cooperate, or conditions unsuitable for HBOT such as angle-closure glaucoma or eustachian tube occlusion.
  3. Unstable vital signs.
  4. Concurrent intracranial hemorrhage, intracranial mass, malignant tumor, uncontrolled epilepsy, psychiatric disorder, coagulation dysfunction, or other severe uncontrolled comorbidities.
  5. Severe pulmonary bullae or emphysema.
  6. Active internal bleeding or coagulopathy.
  7. Uncontrolled hyperpyrexia (body temperature >38.0°C).
  8. Concurrent use of disulfiram, bleomycin, or cisplatin chemotherapy. Relative Contraindications
  9. Uncontrolled hypertension (systolic BP >160 mmHg or diastolic BP >100 mmHg).
  10. Severe cardiac arrhythmias (e.g., third-degree atrioventricular block without a pacemaker, frequent ventricular tachycardia).
  11. Chronic obstructive pulmonary disease (FEV1 <50% of predicted) or active asthma.
  12. Psychiatric or cognitive impairment preventing cooperation with the therapy. Comorbidity Restrictions
  13. End-stage renal disease (dialysis-dependent).
  14. Terminal malignancy (life expectancy <6 months).
  15. Pregnancy or lactation (a negative pregnancy test is required for women of childbearing potential).

      Recent Clinical Events
  16. Acute myocardial infarction or unstable angina within the past 4 weeks.
  17. Hospitalization or emergency department visit for acute heart failure within the past 2 weeks.
  18. Current use of intravenous positive inotropic agents.
  19. Within 6 months after cardiac surgery.
  20. Use of any mechanical circulatory support.
  21. Participants with a 6-minute walk test result exceeding 450 meters or who are unable to complete the test.

      Other Exclusion Conditions
  22. Inability to complete follow-up (e.g., planned relocation, non-compliance with follow-up assessments).
  23. Concurrent participation in any other clinical trial that may interfere with the outcomes of this study.
  24. Unforeseen circumstances judged by the investigators to be ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test | 6MWT will be performed in the experimental group at baseline (pre-HBOT), one day after each HBOT course, and at 3, 6, and 12 months post-treatment.
  The 6MWT is conducted on a 30-meter, flat corridor. Patients walk back and forth as far as possible in 6 minutes. They self-pace and can stop if needed. Standardized encouragement is given. Before and after, vital signs, dyspnea, and fatigue (Borg scale) are recorded. The primary outcome is the total distance walked (6MWD).

SECONDARY OUTCOMES:
Cardiac Color Doppler Ultrasound | Echocardiograms will be performed at baseline, following each HBOT course (1-day), and at 3, 6, and 12-month follow-ups.
  During the test, the patient lies on their left side. A technician places a transducer with gel on the chest to obtain ultrasound images of the heart. It captures real-time images of chamber size, muscle thickness, valve motion, and pumping function (ejection fraction). The procedure is painless, takes about 30-45 minutes, and requires no special preparation.
Cardiopulmonary Exercise Testing (CPET) | CPET will be performed at baseline, 1-day post-each HBOT course, and at 3/6/12-month follow-ups.
  Cardiopulmonary Exercise Testing (CPET) measures how the heart, lungs, and muscles work during exercise. The patient exercises on a treadmill or stationary bike with increasing intensity while wearing a mask to analyze oxygen and carbon dioxide. Vital signs are monitored throughout. The test lasts 10-15 minutes and evaluates overall cardiopulmonary fitness.
Non-Invasive Cardiac Output Monitoring | Non-Invasive Cardiac Output Monitoring (NICOM) results will be recorded at baseline, one day after each hyperbaric oxygen treatment course, and at 3, 6, and 12 months post-treatment.
  Non-Invasive Cardiac Output Monitoring (NICOM) measures heart function without inserting catheters. Electrode sensors are placed on the patient's chest to track blood flow dynamics using bioimpedance or bioreactance technology. The patient remains still during the 10-20 minute test, which provides real-time data on cardiac output and stroke volume. No special preparation is required.
Kansas City Cardiomyopathy Questionnaire | KCCQ will be administered at baseline, 1-day post-each HBOT course, and during 3/6/12-month follow-ups.
  The KCCQ is a self-administered questionnaire. Patients answer 23 items about their heart failure symptoms and how it impacts their life over the past 2 weeks. It takes about 5-10 minutes to complete and produces scores from 0-100, where higher scores indicate better health status and quality of life.
Meta-Analysis Global Group in Chronic Heart Failure | The MAGGIC risk score will be calculated at baseline, one day after each hyperbaric oxygen treatment course, and at 3, 6, and 12 months post-treatment.
  The MAGGIC questionnaire is a 13-item prognostic risk score for heart failure patients. It combines patient data (age, gender, BMI, smoking status) with clinical metrics (ejection fraction, systolic BP, creatinine, NYHA class, medication use) and disease history (diabetes, COPD, heart failure duration). Clinicians collect these parameters to calculate a risk score predicting 1- and 3-year mortality. Completion time is 5 minutes.
Pittsburgh Sleep Quality Index (PSQI) | PSQI will be administered at baseline, 1-day post-each HBOT course, and during 3/6/12-month follow-ups.
  The PSQI is a self-rated questionnaire assessing sleep quality over a 1-month interval. It contains 19 items generating seven component scores: subjective quality, latency, duration, efficiency, disturbances, medication use, and daytime dysfunction. These components yield a global score (0-21), with higher scores indicating worse sleep quality. Administration requires 5-10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No